CLINICAL TRIAL: NCT06442176
Title: Choroid Thickness May Shed Light On Early Coronary Artery Disease
Brief Title: Choroid In Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, ERHAN TENEKECIOGLU, Assoc Prof, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: BSH-131/21
Record Dates: First submitted 2024-05-27; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Choroid Diseases
Keywords: Coronary Artery Disease; Choroid; Gensini Score; Optical Coherence Tomography
MeSH Terms: conditions — Choroid Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Healthy group
  Interventions: Diagnostic Test: OCT
- Coronary Artery Disease Group
  Interventions: Diagnostic Test: OCT

INTERVENTIONS:
Diagnostic Test: OCT — Enhanced depth imaging optical coherence tomography (EDI-OCT) using the Heidelberg Spectralis HRA + OCT (Heidelberg Engineering, Inc., Franklin, MA, USA)

SUMMARY:
Purpose: To investigate any relationship between choroid thickness (CTh) and coronary artery disease (CAD), particularly in its earlier stages before clinically evident.

Design: Retrospective, cross-sectional observational study

Methods:

Setting: The study was performed in two institutions; patients were recruited in Balikesir City Hospital. The ophthalmological examinations and coronary angiograms were performed in Balikesir City Hospital. The analysis of the coronary angiograms including Gensini scoring were conducted in Bursa Education and Research Hospital.

Study Population: The study group comprised 68 patients with documented CAD and 60 healthy control subjects. Patients with high myopia, cataracts, retinal vascular disease, retinal surgery, retinal dystrophy, laser photocoagulation, intravitreal anti-VEGF treatment, glaucoma, uveitis, retinal disorders, any systemic diseases were excluded from the study groups.

Observation Procedure: Refractive examination, corrected visual acuity, intraocular pressure measurements, anterior and posterior segment examinations. Following measurements of macular thickness and retinal nerve fiber layer, choroidal thickness of both eyes was assessed by enhanced depth imaging optical coherence tomography.

ELIGIBILITY:
Inclusion Criteria:

* Normal coronaries at coronary angiography for healthy control group
* Without any coronary artery disease equivalent diseases such as peripheral artery disease, cerebrovascular disease and stroke for healthy control group
* Ability to give informed consent for the study
* Coronary artery disease with stenosis detected in coronary angiogram for coronary artery disease group

Exclusion Criteria:

* High myopia (> 6D)
* Cataracts
* Retinal vascular disease
* Retinal surgery
* Retinal dystrophy
* Laser photocoagulation
* Intravitreal anti-VEGF treatment
* Glaucoma
* Uveitis
* Retinal disorders (comprising diabetic macular edema, diabetic/hypertensive retinopathy, vein occlusions, retinal dystrophy, epiretinal membrane, vitreomacular traction, age-related macular degeneration)
* Any systemic diseases
* Obesity (body-mass index ≥30 kg/m²)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All study participants had coronary angiography performed by the Department of Cardiology on an elective scheduled basis following ischaemic changes detected on treadmill stress test or at least 5% ischaemic burden determined at conventional single-photon emission computed tomography (SPECT) myocardial perfusion imaging (MPI).
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-04-21 (Actual)

PRIMARY OUTCOMES:
Choroidal thickness in Healthy Subjects | 1 day
  micron
Choroidal thickness in patients with coronary artery disease | 1 day
  micron

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Tenekecioglu, MD, Study Director — Balikesir City Hospital; Iskender Kadife, MD, Principal Investigator — Balikesir City Hospital; Erhan Tenekecioglu, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Balikesir City Hospital, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No